CLINICAL TRIAL: NCT05829590
Title: Speech and Image Recognition Based System in Improving Reporting Quality During Colonoscopy
Brief Title: AI-assisted Colonoscopy Report System In Improving Reporting Quality
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Renmin Hospital of Wuhan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: EA-23-002
Record Dates: First submitted 2023-04-02; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-03

CONDITIONS: Artificial Intelligence; Colonoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- with Artificial intelligence assistant system (Experimental): Endoscopists would complete the colonoscopy report with the assistance of the artificial intelligence system.
  Interventions: Diagnostic Test: Artificial intelligence assistant system
- without Artificial intelligence assistant system (No Intervention): Endoscopists would complete the colonoscopy report without special prompts.

INTERVENTIONS:
Diagnostic Test: Artificial intelligence assistant system — The artificial intelligence assistant system can automatically capture bowel segment images and prompt abnormal lesions based on speech recognition and deep learning.
  Arms: with Artificial intelligence assistant system

SUMMARY:
In this study, the investigators proposed a prospective study about the effectiveness of speech and image recognition-based system in improving reporting quality during colonoscopy for colonoscopy report quality in endoscopists. The participants would be divided into two groups. For the collected colonoscopy videos, group A would record their observations with the assistance of the artificial intelligence system. The artificial intelligence assistant system can automatically capture bowel segment images and prompt abnormal lesions. Group B would complete the endoscopy report without special prompts. After a period of washout period, the two groups switched, that is, group A without AI assistance and group B with AI assistance to complete the colonoscopy report. Then, the completeness of the colonoscopy report, the completeness of capturing anatomical landmarks and detected lesions, the completeness of structured description, the accuracy of lesion reporting, the time for reporting and the satisfaction with the reporting system are compared with or without AI assistance.

ELIGIBILITY:
Inclusion Criteria:

Patients:

1. Male or female ≥18 years old;
2. Able to read, understand and sign an informed consent;
3. The investigator believes that the subjects can understand the process of the clinical study, are willing and able to complete all study procedures and follow-up visits, and cooperate with the study procedures;
4. Patients requiring colonoscopy.

Doctors:

1. Males or females who are over 18 years old;
2. After qualified medical education and obtaining the Physician's Practice License.

Exclusion Criteria:

Patients:

1. Have drug or alcohol abuse or mental disorder in the last 5 years;
2. Pregnant or lactating women;
3. Patients with known multiple polyp syndrome;
4. patients with known inflammatory bowel disease;
5. known intestinal stenosis or space-occupying tumor;
6. known colon obstruction or perforation;
7. patients with a history of colorectal surgery;
8. Patients with a previous history of allergy to pre-used spasmolysis;
9. Unable to perform biopsy due to coagulation disorders or oral anticoagulants;
10. High-risk diseases or other special conditions that the investigator considers the subject unsuitable for participation in the clinical trial.

Doctors:

1. The researcher believes that the subjects are not suitable for participating in clinical trials.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-06-15 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The integrity of colonoscopy report | One month
  Report integrity with or without AI-assisted. Calculation method = number of information recorded / total number of information need to record x 100%

SECONDARY OUTCOMES:
The integrity of capturing anatomical landmarks | One month
  The integrity in captured bowel landmrak images with or without AI-assisted. Calculation method = number of anatomical landmarks in captured images / total number of anatomical landmarks x 100%

OTHER OUTCOMES:
The integrity of report lesion | One month
  Report lesion integrity with or without AI-assisted. Calculation method = number of report lesions / total number of lesions x 100%
The completeness of structured description | One month
  The completeness of structured description with or without AI-assisted. Calculation method = number of structured descriptions / total number of structured descriptions need to record x 100%
Accuracy of lesion reporting | One month
  Accuracy of lesion report with or without AI-assisted. Calculation method = number of lesions with correct description / total number of lesions descriptionx 100%
The time for reporting | One month
  The time for reporting with or without AI-assisted
The satisfaction with the reporting system | One month
  The satisfaction with the reporting system with or without AI-assisted

CONTACTS AND LOCATIONS:
Locations (1):
- Renmin Hospital of Wuhan Univercity, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No